CLINICAL TRIAL: NCT01939015
Title: 3D Vs Standard Miniplate in Fixation of the MAFs
Brief Title: Three Dimensional Versus Standard Miniplate In Fixation Of Mandibular Angle Fracture- A Prospective Randomized Controlled Clinical Trial
Acronym: RCTs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Thamar University (Other)
Responsible Party: Principal Investigator, ESSAM ALMORAISSI, lecturer in Faculty of Dentistry,Dhamar University,Yemen, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201301; OMFS201301 (Other: faculty of oral and dental medicine,Cairo univeristy)
Record Dates: First submitted 2013-08-22; First posted 2013-09-11 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Displaced Mandibular Angle Fracture
Keywords: 3D miniplate; angle mandibular fracture; champy technique; internal rigid fixation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard titanium miniplate- single non compression miniplate (Active Comparator): fixation will be perform by A single non compression miniplate with 4-hole 2-mm using 2-mm monocortical screws at superior border of the mandible according to ideal lines of osteosynthesis.
  Interventions: Device: 3D titanium miniplate; Device: Standard titanium miniplate- single non compression miniplate
- three dimensional titanium miniplate (Experimental): 3D curved strut miniplate* (Universal Mandible System, Stryker-Lei binger, Freiburg, Germany) , installed and stabilized with monocortical screws. The 3D plate will be place in such a way that a horizontal bar is perpendicular and a vertical bar is parallel to the fracture line.
  Interventions: Device: 3D titanium miniplate; Device: Standard titanium miniplate- single non compression miniplate

INTERVENTIONS:
Device: 3D titanium miniplate — for study group by using 3D titanium miniplate under open reduction under general anesthesia with mono cortical screw, while in control group single titanium miniplate at superior border with mono cortical screw according to ideal line of osteosynthesis of champy
  Other Names: Universal Mandible System, Stryker-Lei binger, Freiburg, Germany
Device: Standard titanium miniplate- single non compression miniplate — single non compression miniplate placed at superior border with monocortical screws via intraoral approach
  Other Names: Champy technique (single non compression miniplate)

SUMMARY:
* The aim of this study is to compare the standard and 3D miniplates fixation in mandibular angle fractures regarding to wound dehiscence, infection, nonunion, pain, hypoesthesia, and malocclusion. and to analyze advantages and disadvantages of one method over the other.
* Radiographic follow-up (in the form of posteroanterior and panoramic radiographs) will used to evaluate the patients immediately and 2 and 4 months postoperatively. Patients returned 7 days after surgery for clinical evaluation . The patients will be examined radiographically for accuracy of the reduction, screw positioning, adverse reactions in the vicinity of screw placement, and bone healing. the complications encountered will be recorded and treated. The clinical evaluations will be performed by 1 surgeon at each institution.
* The patients will also evaluated clinically for infection, nonunion, pain, hypoesthesia, and malocclusion. Malocclusion will assessed based on patient complaints. Criteria for infection will based on either of the following conditions: 1) purulent discharge from an incision and 2) serosanguineous drainage and a wound culture positive for a known pathogen. All the patients will evaluated postoperatively by a single assessor.
* Statically analysis :

Student's t test will be used to compare 3D and Champy's miniplate fixation. A value of P ≤ 0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
* This study will include 20 dentate patients with mandibular angle fracture whom presented for treatment at Department Of Oral and Maxillofacial Surgery, Faculty Of Oral And Dental Medicine, Cairo University.
* The patients after inclusion will be randomly divided into either Group A or Group B. Group A consist of 10 patients underwent open reduction with internal fixation of the angle mandibular fracture with 3D titanium miniplates whereas Group B consist of 10 patients underwent open reduction with internal fixation of the mandibular angle fracture with standard miniplate using a single miniplate technique of Champy's principle of osteosynthesis.
* Inclusion criteria: 1) Age group between 15-40 years. 2) patients with non-infected and non-comminuted mandibular angle fractures 3) surgical treatment provided within 7 days of injury via open reduction and internal fixation (ORIF) by an extra oral approach 4) no use of postsurgical maxillomandibular fixation (MMF) postoperatively 5) a 1-week duration of postsurgical oral antibiotic therapy.
* Exclusion criteria : 1) the fracture was infected at the time of treatment, 2) medical conditions that could possibly have interfered with healing (diabetes, chemotherapy, etc.) or prevented general anesthesia.
* Preoperative Evaluation

Careful extra and intraoral clinical examinations will be perform on all patients. The presence of lacerations, swelling, ecchymosis, occlusal disturbances, or broken, avulsed, or missing teeth will noted, and the mandibular movements, maximal interincisal opening, and nerve function will be recorded. Palpation of the mandible for areas of tenderness, segment mobility, bony crepitus, and tooth mobility will be also perform . Radiographic images (panoramic and posteroanterior) will be taken to evaluate the fracture. Immediately preoperatively, each patient will be given a standard dose of 1.5 g of Unasyn* and 8 mg of Epidron** intravenously.

-Surgical Technique:

After placement of arch bars, the fracture line will be exposed through extraoral a submandibular (Risdon) incision. Only the amount of soft tissue stripping necessary to visualize, reduce, and stabilize the fracture will be performed. Mobile teeth or teeth with apices that will be exposed in the fracture will be removed.

All a fracture site will be identified, reduced, and after obtaining satisfactory occlusion, temporary maxillomandibular fixation will be placed using either Erich's arch bar or Ivy loop eyelet wiring.

Fixation in group A will be achieved using a 3D curved strut miniplate* (Fig 1) , installed and stabilized with monocortical screws. The 3D plate will be place in such a way that a horizontal bar is perpendicular and a vertical bar is parallel to the fracture line. While in group B fixation will be perform by A single non compression miniplate with 4-hole 2-mm using 2-mm monocortical screws.

In both group fixation will be carried out through extraoral submandibular approach and placed in the neutral zone of the mandibular angle (between tension and compression areas).

After fixation of the fracture, intermaxillary fixation will be removed . And the incisions will be close in layers by absorbable suture while the skin closed by 5-0 nylon sutures. No drains will placed. and the occlusion will checked .

-Postsurgical Management:

Antibiotics will be continued through the preoperative period and for 5 to 7 days after surgery. And other medication to control swelling and pain will be administered. Chlorhexidine mouth rinse will be provided for all patient until removal of arch bars. Soft diet will be strongly recommend for 2 weeks then Pasty diet will be gradually regained .

-Postoperative Evaluation :

Radiographic follow-up (in the form of posteroanterior and panoramic radiographs) will used to evaluate the patients immediately and 2 and 4 months postoperatively. Patients returned 7 days after surgery for clinical evaluation . The patients will be examined radiographically for accuracy of the reduction, screw positioning, adverse reactions in the vicinity of screw placement, and bone healing. the complications encountered will be recorded by treatment scoring system and treated. The clinical evaluations will be performed by 1 surgeon at each institution.

The patients will also evaluated clinically for infection, nonunion, pain, hypoesthesia, and malocclusion. Malocclusion will assessed based on patient complaints. Criteria for infection will based on either of the following conditions: 1) purulent discharge from an incision and 2) serosanguineous drainage and a wound culture positive for a known pathogen. All the patients will evaluated postoperatively by a single assessor.

-Statically analysis :

Student's t test will be used to compare 3D and Champy's miniplate fixation. A value of P ≤ 0.05 will be considered statistically significant.

ELIGIBILITY:
* Inclusion Criteria:

  * Adults dentate patients (>17 years old) with displaced an angle mandibular fracture
  * non infected non comminuted angle mandibular fracture
* Exclusion Criteria:

  * infected angle mandibular fracture
  * atrophied mandibular fracture
  * angle fracture with subcondylar fracture
  * patients under 17 year
  * gun shout injury associated fracture

Ages: 17 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 6 monuths
  1. Wound dehiscence (binary outcome) by Clinical examination
  2. mal /un union (binary outcome) by Clinical examination
  3. Evaluation of Occlusion (binary outcome) (Only after 3 months of fracture treatment) by using the treatment scoring system35 Surgeon's evaluation
     * 5 points: occlusion altered bilaterally. Reoperation required.
     * 3 points: occlusion altered on one side: Reoperation required
       * 1 point: occlusion altered on one side. The other side has to be adjusted.
       * 3 points: occlusion adequate on both sides but not the same as before injury.
       * 5 points: occlusion the same as before injury.

SECONDARY OUTCOMES:
Radiographic follow-up | 6 months
  The patients will be examined radiographically for accuracy of the reduction, screw positioning, adverse reactions in the vicinity of screw placement, and bone healing by using digora software.

OTHER OUTCOMES:
mouth opening | 7 days
  BY USING BOELY GAUGE IN MILLIMTER

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial SurgeryFaculty of Oral and Dental Medicine, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Derived] Al-Moraissi EA, Mounair RM, El-Sharkawy TM, El-Ghareeb TI. Comparison between three-dimensional and standard miniplates in the management of mandibular angle fractures: a prospective, randomized, double-blind, controlled clinical study. Int J Oral Maxillofac Surg. 2015 Mar;44(3):316-21. doi: 10.1016/j.ijom.2014.10.012. Epub 2014 Nov 15. PMID 25457871